CLINICAL TRIAL: NCT00676611
Title: Both Column Acetabular Fractures With Associated Posterior Deformity Patterns: Implications for Surgical Treatment and Prognosis
Brief Title: Acetabular Fractures of Both Columns
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: DCG001; IRB# 27556EP
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Acetabular Fractures; Both Columns
Keywords: Acetabular Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to study a specific acetabular (hip socket) fracture pattern and how its treatment affects the functional, clinical, and x-ray outcomes. There are no experimental procedures involved.

DETAILED DESCRIPTION:
This study will identify a small subset of patients that fall outside the Letournel classification system of acetabular fractures. The fracture pattern, its influence on the surgical treatment decision making process, and the radiographic and outcomes will be detailed. In particular, both-column acetabular fractures with significant posterior deformity have been correlated with poor functional outcomes, increased arthritis radiographically, and worse prognosis in general. Despite these findings, there has been no specific study evaluating these injury patterns to date. We present ten patients with both column acetabular fractures and an associated posterior column/wall piece and their clinical outcomes in an effort to help guide surgical treatment and offer prognostic guidance.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent surgical fixation of the hip at Hershey Medical Center between June 2006 and May 2007 by Dr's J. Spence Reid and David Goodspeed.
* They will include patients that are admitted directly from the field or are transferred from outside hospitals.

Exclusion Criteria:

* will be those acetabular fractures of non-traumatic etiology (e.g.: secondary to malignancy or fatigue)
* fractures that have not undergone operative fixation
* pediatric populations under the age of 18
* mentally compromised patients
* those that do not give consent for the clinical evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 10 patients who have had column fractures with an associated posterior wall fracture or significantly displaced posterior column fracture that required a separate approach for reduction and/or fixation of the hip performed at Hershey Medical Center by two surgeons, Drs. David Goodspeed and J. Spence Reid over a 12 month period (June 2006 - May 2007). There is no control population.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-05; Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Goodspeed, MD, Principal Investigator — Penn State Milton S. Hershey
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States